CLINICAL TRIAL: NCT06465277
Title: Assessment of Right Ventricular Contractile Reserve Following Lung Resection by Dobutamine Stress Cardiac Magnetic Resonance: a Feasibility Study
Brief Title: CMR Right Ventricular Contractile Reserve Following Lung Resection
Status: Recruiting | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22066JS-AS
Record Dates: First submitted 2023-09-06; First posted 2024-06-18 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Surgery; Anesthesia
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples frozen for batch analysis of cardiac biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Lung resection: 12 patients undergoing lobectomy. Pre and post-operative dobutamine stress CMR testing and cardiac biomarker testing.
  Interventions: Diagnostic Test: Dobutamine stress CMR; Diagnostic Test: Cardiac biomarker sample
- Oesophagectomy: 15 patients Peri-operative cardiac biomarker testing.
  Interventions: Diagnostic Test: Cardiac biomarker sample
- Gastrectomy: 15 patients Peri-operative cardiac biomarker testing.
  Interventions: Diagnostic Test: Cardiac biomarker sample

INTERVENTIONS:
Diagnostic Test: Dobutamine stress CMR — Dobutamine stress testing will be undertaken in keeping with local departmental clinical guidelines with a graded increase in dobutamine infusion up to a maximum of 10microgram/kg/min. The patients' medications will be managed in keeping with the usual clinical practice and departmental guidelines.
  At rest and on each graded level of dobutamine infusion we will collect cine loops of the cardiac cycle including a short-axis stack of the ventricles, a four-chamber view and flow imaging perpendicular to the main, left and right pulmonary arteries.
  Post-processing will be dual reported by blinded observers using the Argus analysis software (Siemens) according to a standardised protocol. A safety report of each CMR scan will be generated by a consultant cardiologist, any abnormalities identified will be referred to the appropriate medical speciality and highlighted to the patient's clinical team.
  Groups: Lung resection
Diagnostic Test: Cardiac biomarker sample — blood samples will be collected pre-operatively, in recovery, on post-operative days 1 and 2, and at 4-8 weeks post-operatively

SUMMARY:
Feasibility study investigating CMR dobutamine stress testing before and after lung resection

DETAILED DESCRIPTION:
We hypothesise that following lung resection,

1. the subtle decrease in RV function and increase in afterload we have demonstrated at rest is associated with a marked impairment of RV function on exercise, termed impaired RV contractile reserve (RVCreserve),
2. impaired RVCreserve is associated with impaired functional capacity .

In this study we aim to assess the feasibility of dobutamine stress cardiovascular magnetic resonance (CMR) scanning to assess RVCreserve pre- and post-operatively in patients undergoing lung resection.

Additionally, we hypothesise that one lung ventilation (with and without lung resection) is associated with biomarker evidence of RV injury.We will perform peri-operative cardiac biomarkers to differentiate between the contribution of major surgery (gastrectomy, lung resection and oesophagectomy), one lung ventilation (lung resection and oesophagectomy) and lung resection on RV injury.

ELIGIBILITY:
Inclusion Criteria:

* 1) Provision of informed consent 2) Age >16 years 3) Planned elective

  1. lobectomy lung resection or
  2. oesophagectomy surgery with one lung ventilation or
  3. gastrectomy

Exclusion Criteria:

1. Pregnancy
2. On-going participation in any investigational research which could undermine the scientific basis of the study
3. Atrial fibrillation at baseline
4. Any contraindication to

   a. CMR, i. Cardiac pacemaker, artificial heart valve, neurostimulator, cochlear implant ii. Aneurysm clips iii. Metal injuries to the eye iv. Loose metal in a part of the body b. Dobutamine stress testing as per the Society for Cardiovascular Magnetic Resonance64 i. Severe systemic arterial hypertension (≥220/120 mmHg) ii. Unstable angina pectoris iii. Severe aortic valve stenosis (peak aortic valve gradient >60mmHg or aortic valve area < 1cm2) iv. Complex cardiac arrhythmias including uncontrolled atrial fibrillation v. Hypertrophic obstructive cardiomyopathy vi. Myocarditis, endocarditis, or pericarditis vii. Uncontrolled heart failure
5. Lung resection specific

   1. Wedge, segmental or sub-lobar lung resection
   2. Pneumonectomy
   3. Isolated right middle lobectomy

      -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting for surgical resection of lung, oesophagus or stomach.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1) Feasibility of dobutamine stress CMR to measure RVCreserve following lung resection. | Pre-operative and 2 months post-operative
  Reliability and variability will be assessed through dual reporting of the CMR images, testing intra-/inter-observer intraclass correlation coefficient (ICC) and coefficient of variation (CV). Study design will allow comparison to our previous resting studies published exercise literature and between pre- and post-operative imaging.

SECONDARY OUTCOMES:
1) Acceptability of the dobutamine stress CMR protocol to patients, by questionnaire | Pre-operative and 2 months post-operative
  Assessed by patient satisfaction questionnaires rate compared to our previous CMR studies that were performed without dobutamine stress testing.
1) Acceptability of the dobutamine stress CMR protocol to patients, by completion | Pre-operative and 2 months post-operative
  Assessed by patient recruitment/withdrawal rate compared to our previous CMR studies that were performed without dobutamine stress testing.
2) Incidence of complications related to dobutamine stress CMR | Pre-operative and 2 months post-operative
  We will assess for the onset of any of the following during the scan
  1. New onset atrial fibrillation
  2. Ventricular tachycardia
  3. Angina, chest pain, shortness of breath and/or ischaemic ECG changes
3) Change in RVCreserve change following lung resection | Pre-operative and 2 months post-operative
  Comparison of the change in RVEF on stress pre- and post-operatively
4) Change in PVreserve change following lung resection | Pre-operative and 2 months post-operative
  Comparison of change in wave reflection on stress pre- and post-operatively
5) Association between the changes in RVCreserve and markers of cardiac inflammation, BNP | Pre-operative and 2 months post-operative
  Comparison of change in RVCreserve and the change in BNP
5) Association between the changes in RVCreserve and markers of cardiac inflammation, hsTnT | Pre-operative and 2 months post-operative
  Comparison of change in RVCreserve and the change in hsTnT.
1) Post-operative change in BNP | Peri-operative blood samples, pre-op, immediately post-op, post-op days 1 and 2, 4-8 weeks post-op
  Post-operative change in BNP in oesophagectomy compared to lung resection and gastrectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Belfast Health and Social Care Trust, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No